CLINICAL TRIAL: NCT06748274
Title: The Brain-heart-gut Connection (BHG-CONNECT): Targeting the Frontal-vagal Pathway to Personalize Noninvasive Brain Stimulation
Brief Title: The Brain-Heart-Gut Connection
Acronym: BHG-CONNECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: Medical School Berlin (Other); Universitäre Psychiatrische Dienste Bern (UPD), Switzerland (Unknown)
Responsible Party: Principal Investigator, Jessica Jacobs, PhD Candidate, University of Bern
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BHG-CONNECT; 2024-D0080 (Other: Kantonale Ethik Kommission (KEK) Bern)
Record Dates: First submitted 2024-12-10; First posted 2024-12-27 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Major Depression; Functional Dyspepsia; Autonomous Dysfunction
Keywords: Depression; Brain-Heart Coupling; Brain-Gut Axis; Non-invasive Brain Stimulation; TMS; tDCS; Functional dyspepsia; Connectivity
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: For this bicentric (Bern and Berlin), cross-over, single-blind, controlled trial with partial randomization, we will recruit n=32 healthy participants (Study Arm 1, Bern and Berlin) and n=32 participants expressing predefined elevated scores in depressive and autonomic symptoms, including functional dyspepsia (Study Arm 2, Bern). Notably, sample sizes of Study Arms 1 and 2 are estimates and will be adjusted using Bayesian updating (see "Power considerations and key analysis plan"). Before starting any of the study arms, n=10 participants (n=5 in Bern, n=5 in Berlin) will be invited to undergo the protocol for Study Arm 1 to ensure technical feasibility and high data quality (Pilot Phase).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants will be held uninformed about the interventional condition undertaking. TMS will be single-blinded, as the stimulation is applied over three active control spots, while tDCS will be double-blinded, with protocols initiated remotely.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Frontal Mapping (Other): To identify the individual TMS stimulation spot and intensity, the Heart-Brain Coupling protocols described by Dijkstra and colleagues (2023) are applied over 8 different spots. To identify the individual stimulation intensity, trains of 10 Hz for 5 seconds with an inter-train interval of 11 seconds are applied (Dash protocol). The subjects are stimulated with 15 different intensities, raising in 2% machine output steps. The starting intensity is set as 28% below the motor threshold (MT), leading to the highest intensity level of 120% MT at step 15. The intensity causing the HR to decelerate the most will be taken as the individual stimulation intensity for subsequent sessions.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- TMS - Grid-spot (Experimental): Subjects receive active rTMS over the individual DLPFC spot. Both sessions follow the same protocol and procedures. The 10Hz Dash protocol is applied for about 18.75minutes with the individual intensity defined in the frontal mapping session (arm 1).
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- TMS control (Cz) (Active Comparator): Subjects receive active TMS over the central midline. Both sessions follow the same protocol and procedures. The rTMS 10 Hz Dash protocol is applied for about 18.75 minutes with the individual intensity defined in the frontal mapping session (arm 1)
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- HD-tDCS (anodal) (Experimental): Subjects receive anodal tDCS over the personalized stipulation spot (arm 1) for a total of 18.75 minutes with an intensity of 2mA.
  Interventions: Device: High-definition transcranial direct current stimulation (HD-tDCS)
- HD-tDCS control (cathodal) (Active Comparator): Subjects receive cathodal tDCS over the personalized stimulation spot (arm 1) for a total of 18.75 minutes with an intensity of 2mA.
  Interventions: Device: High-definition transcranial direct current stimulation (HD-tDCS)
- rTMS - Beam F3 (Active Comparator): Subjects receive active TMS over the Beam-F3 spot. All 3 TMS sessions follow the same protocol and procedures. The rTMS 10 Hz Dash protocol is applied for about 18.75 minutes with the individual intensity defined in the frontal mapping session (arm 1).
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — Transcranial Magnetic Stimulation (TMS) is a sophisticated neuromodulation technique that involves the use of a magnetic coil placed against the scalp to generate brief magnetic pulses. These pulses induce electric currents in the cortical neurons, leading to depolarization or hyperpolarization depending on the parameters of the stimulation.
  Arms: Frontal Mapping; TMS - Grid-spot; TMS control (Cz); rTMS - Beam F3
Device: High-definition transcranial direct current stimulation (HD-tDCS) — Transcranial Direct Current Stimulation (tDCS) is a non-invasive brain stimulation technique that involves applying a low-intensity electrical current to specific areas of the scalp. The electric current induces alterations in the membrane potentials of underlying neuronal networks. The application of tDCS with concentric ring electrodes is a more targeted form of tDCS, allowing for more precise modulation of cortical activity compared to traditional tDCS methods.
  Arms: HD-tDCS (anodal); HD-tDCS control (cathodal)

SUMMARY:
Major Depressive Disorder (MDD) often co-occurs with cardiovascular and gastrointestinal symptoms, highlighting the importance of the brain-heart-gut connection in developing comprehensive treatments. Previous research suggests that key hubs in the depression network, such as the dorsolateral prefrontal cortex (DLPFC) and the subgenual anterior cingulate cortex (sgACC), overlap with structures that are involved in autonomic control, particularly the vagus nerve. Repetitive transcranial magnetic stimulation (rTMS) to the left DLPFC is an established treatment for MDD; however, antidepressant efficacy varies greatly across individuals, and optimal DLPFC targeting remains a significant challenge. Personalized rTMS based on DLPFC-sgACC connectivity improves outcomes but is limited by practical and financial constraints. Recently, rTMS-induced heart-brain coupling (HBC) has emerged as a promising method to utilize heart rate responses to guide treatment. The primary goal of this project is to personalize HBC to improve DLPFC-based targeting for the treatment of MDD while also probing additional readouts of the frontal-vagal system. In Study Arm 1, we will implement an innovative frontal mapping technique to identify the personalized "Grid-Spot" that elicits the strongest HBC in healthy participants. In subsequent visits, we will compare heart rate responses during the 10Hz "Dash" protocol between the "Grid-Spot", conventional DLPFC targeting using "Beam-F3" and an active control region (Cz). Additionally, we will integrate various autonomic nervous system (ANS) measures, including gut motility, pupil dilation and electrodermal activity (EDA), to explore the brain-heart-gut axis and assess their utility in improving target engagement. Furthermore, we will extend our methodology to the personalized application of high-definition transcranial direct current stimulation (HD-tDCS). Specifically, we will explore the effects of anodal versus sham HD-tDCS over the HBC-guided "Grid-Spot" on ANS readouts and compare these outcomes to those observed with rTMS. In Study Arm 2, we will repeat experimental rTMS visits from Study Arm 1 with participants exhibiting elevated symptom scores in depression, autonomic dysfunction and functional dyspepsia. In Study Arm 2 we will also validate our optimal "Grid-Spot" identification through neuroimaging of DLPFC-sgACC connectivity. This project will deepen our understanding of the brain-heart-gut connection and contribute to more accessible, personalized brain stimulation treatments for MDD.

DETAILED DESCRIPTION:
Major Depressive Disorder is estimated to affect 5% of the global population, which makes it the most common mental disorder in the world. It is well-established that it is associated with abnormal autonomic nervous system function. Commonly co-occurring symptoms such as increased heart rate, reduced heart rate variability, or gastric hypomotility suggest a complex interplay of pathological brain networks and autonomic regulation. Notably, individuals with depression face a higher likelihood of developing cardiovascular disease, whereas individuals with cardiovascular diseases have a higher probability of developing depression. Gastrointestinal symptoms such as delayed gastric emptying, diarrhea, or abdominal pain are found significantly more often in depressed compared to non-depressed individuals. Therefore, a deeper understanding of the brain-heart-gut connection is crucial for developing more comprehensive and effective treatment strategies.

The frontal-vagal network theory offers a neuroanatomical framework for understanding the comorbidity of cardiovascular and gastrointestinal diseases in depression. The theory states that major hubs of the depression network, such as the dorsolateral prefrontal cortex and the subgenual anterior cingulate, overlap with structures that are involved in autonomic control, particularly the vagus nerve. Stimulation of these areas using neuromodulation therapies such as repetitive transcranial magnetic stimulation, deep brain stimulation, or vagus nerve stimulation has been linked to symptom improvement. Interestingly, vagus nerve stimulation has also been identified as a potential therapy for cardiovascular disorders, such as cardiac arrest and stroke. Furthermore, recent studies demonstrate promising results in applying transcutaneous auricular vagus nerve stimulation to treat functional dyspepsia, a common functional gastrointestinal disorder characterized by altered motility, which contributes to symptoms such as postprandial fullness, early satiation, epigastric pain, and burning.

The left dorsolateral prefrontal cortex is the most accessible and most used target within the frontal-vagal network for applying repetitive transcranial magnetic stimulation in depression treatment. However, the antidepressant efficacy of repetitive transcranial magnetic stimulation varies significantly between individuals and may depend on the exact stimulation location. To localize the left dorsolateral prefrontal cortex, clinicians often rely on head measurements, such as the '5 cm rule' or the 'Beam-F3 method.' While the '5 cm rule' identifies the left dorsolateral prefrontal cortex as being 5 cm anterior to the motor hotspot, the 'Beam-F3 method' is based on the 10-20 electroencephalography system to account for differences in head dimensions. Software has been developed to estimate the F3 electrode position based on a few head measurements. Both methods are cost-efficient but are not reliable in localizing the optimal left dorsolateral prefrontal cortex stimulation site. More importantly, repetitive transcranial magnetic stimulation has been conceptualized as a depression network therapy. Although stimulation is commonly applied to the left dorsolateral prefrontal cortex, its effects are mediated via distributed networks. In fact, it has been shown that functional connectivity between the left dorsolateral prefrontal cortex and the subgenual anterior cingulate predicts antidepressant response robustly. More specifically, dorsolateral prefrontal cortex stimulation sites with better clinical efficacy were more negatively correlated (anticorrelated) with the subgenual anterior cingulate. Therefore, repetitive transcranial magnetic stimulation personalization based on individual anticorrelation patterns is highly recommended and gained importance with the recent clearance of Stanford Neuromodulation Therapy, an accelerated intermitted theta burst stimulation protocol with functional-connectivity-guided targeting. However, practical and financial challenges constrain the feasibility of utilizing functional magnetic resonance imaging-derived connectivity data in clinical practice.

Based on these considerations, the authors' collaborator and his group have recently proposed a novel approach for guiding stratified transcranial magnetic stimulation treatment of depression. The so-called neurocardiac-guided transcranial magnetic stimulation requires the use of heart rate monitoring during prefrontal repetitive transcranial magnetic stimulation to measure heart rate deceleration as an index of frontal-vagal activation. Several studies were able to replicate this effect in healthy as well as in depressed individuals. Even more recently, the method of neurocardiac-guided transcranial magnetic stimulation evolved through an investigation focusing on the entrainment of the cardiac rhythm as a function of transcranial magnetic stimulation cycle time, the so-called heart-brain coupling. It is hypothesized that stimulation results in bradycardia, whereas the subsequent rest period allows normalization of heart rate, leading to a specific rhythm depending on stimulation parameters. Repetitive transcranial magnetic stimulation-induced heart-brain coupling was validated for the 10 Hz Dash protocol, which shortens the inter-train interval to 11 seconds, enabling faster delivery of stimulation trains without losing efficacy. Notably, the protocol was cleared in 2016, allowing for more convenient depression treatment sessions with a reduced duration of 18.75 minutes. Heart-brain coupling assessed during the Dash protocol has been used for site selection (left versus right) and to determine which of the two commonly used targets ('5 cm rule' versus 'Beam-F3 method') is more effective, indicating that Beam-F3 leads to a stronger frontal-vagal involvement. In addition, this method allows measuring the 'frontal excitability threshold,' defined as the lowest intensity needed to induce heart-brain coupling and therefore recommended to effectively stimulate the dorsolateral prefrontal cortex. Importantly, neuroimaging data supports the underlying role of the prefrontal-subgenual pathway showing maximal heart-brain coupling at dorsolateral prefrontal cortex sites that were anti-correlated with the subgenual anterior cingulate. Thus, repetitive transcranial magnetic stimulation-induced heart-brain coupling has shown the potential to stratify individuals to dorsolateral prefrontal cortex targets with negative subgenual anterior cingulate connectivity and may serve as a biomarker for target engagement with non-invasive brain stimulation. However, the heart-brain coupling protocol currently only enables stratification between dorsolateral prefrontal cortex targets according to the '5 cm rule' and the 'Beam-F3 method,' potentially overlooking the optimal stimulation site based on the strongest negative subgenual anterior cingulate connectivity. This underscores the need to incorporate personalized targets into this approach.

As a cost-effective and easily accessible alternative to transcranial magnetic stimulation, high-definition transcranial direct current stimulation could also be enhanced through personalized targeting via heart-brain coupling. Similar to conventional transcranial direct current stimulation, high-definition transcranial direct current stimulation can facilitate or inhibit the neuronal excitability in the target area, based on the polarity of the center electrode in relation to the surrounding electrodes. To date, there is little knowledge about the link of high-definition transcranial direct current stimulation to autonomic function and the frontal-vagal pathway. In contrast to transcranial magnetic stimulation, transcranial direct current stimulation does not induce action potentials but shifts the resting membrane potential, which in turn influences the firing pattern of the neuronal networks. However, a study showed that the application of anodal high-definition transcranial direct current stimulation over the dorsolateral prefrontal cortex induced modulation of heart rate and heart rate variability in healthy subjects. Additionally, anodal transcranial direct current stimulation of the left dorsolateral prefrontal cortex was found to enhance vagus nerve activity compared to sham stimulation. These findings indicate that transcranial direct current stimulation over the dorsolateral prefrontal cortex activates the frontal-vagal pathway, causing effects comparable to transcranial magnetic stimulation. Therefore, incorporating the heart-brain coupling protocol to personalize high-definition transcranial direct current stimulation targeting could lead to stronger stimulation effects.

The principle of heart-brain coupling serves as a foundation for further exploring the frontal-vagal pathway and potential additional biomarkers that can indicate target engagement. Since the vagus nerve is involved in all parasympathetic functions, stimulation of the frontal-vagal pathway might also have beneficial effects on other autonomic nervous system functions. Given the notably high comorbidity of depression and gastrointestinal symptoms and disorders such as functional dyspepsia, another focus of this proposal lays on stimulation effects on the frontal-vagal pathway in the gastrointestinal tract.

The gut-brain axis represents a complex, bidirectional communication network including the vagus nerve that connects the brain and the gastrointestinal tract and plays a key role in the pathophysiology of both gastrointestinal and psychiatric disorders. Notably, approximately one-third of patients with functional dyspepsia show decreased activity in vagal efferents, which transmit signals from the brain to the gut. Consistent with this, transcutaneous auricular vagus nerve stimulation has been shown to improve functional dyspepsia by enhancing vagal efferent activity and gastric motility as measured with electrogastrogram. Additionally, recent research demonstrated that transcranial magnetic stimulation could alleviate intestinal discomfort in patients with functional bowel disease, another common gastrointestinal disorder characterized by dysmotility and secretion issues. These findings suggest that understanding and intervening in the brain-gut axis by stimulating the frontal-vagal network offers a promising pathway for therapeutic advancements in both gastrointestinal and psychiatric disorders.

Another interesting parameter for exploring the frontal-vagal pathway is heart rate variability. Heart rate variability encompasses two key aspects: heart rate and its variability, reflecting the complex interplay between sympathetic and parasympathetic nervous system influences. Increased vagal tone is associated with heart rate deceleration and heightened heart rate variability, which are indicators of better adaptability and stress resilience. In line, patients with depression express a reduced heart rate variability. Several studies have investigated the effects of non-invasive brain stimulation on heart rate and heart rate variability. A meta-analysis has reported that repetitive transcranial magnetic stimulation applied to prefrontal areas is effective in decreasing heart rate and increasing heart rate variability with larger effects in transcranial magnetic stimulation as compared to transcranial direct current stimulation. Therefore, recording heart rate variability while stimulating could derive valuable insights into its effects on autonomic regulation and might be used as an additional readout of target engagement.

Probably the most promising parameter for an immediate readout of target engagement is pupil dilation, which is defined by the iris dilator muscle (sympathetic control) and the iris sphincter muscle (parasympathetic control). Non-luminance-mediated changes in pupil diameter have a long history of being utilized as a fast and easy-to-access measure of autonomic modulation. There is evidence connecting pupil size with the activity of the norepinephrine-containing neurons in the brainstem nucleus locus coeruleus. Interestingly, the locus coeruleus seems to be associated with two hubs of the frontal-vagal network; the anterior cingulate cortex and the vagus nerve. Vagus nerve stimulation seems to activate the locus coeruleus noradrenergic system, which is altering pupil size. Based on this, targeted dorsolateral prefrontal cortex stimulation might have an instant influence on pupil dilation mediated by the induced change of vagal activity.

Electrodermal activity is another potentially useful parameter, which is primarily controlled by the autonomic nervous system, particularly its sympathetic branch. Electrodermal activity varies depending on the psychophysiological state of the individual and is commonly used as an indicator of emotional and physiological arousal. As the dorsolateral prefrontal cortex is stimulated, changes in sympathetic outflow could lead to variations in electrodermal activity, reflecting alterations in physiological arousal and autonomic function. Physiological responses provide the possibility to observe psychological changes in real-time. Therefore, monitoring electrodermal activity during non-invasive brain stimulation might provide valuable insights into the engagement of the targeted neural pathways.

ELIGIBILITY:
In study arm 1, all participants are healthy between 18 and 65 years of age, and able to give written informed consent.

In study arm 2, all participants must be between 18 and 65 years of age and additionally fulfill the following criteria:

* Elevated autonomic symptom score (> 20) on the Composite Autonomic Symptom Score
* Depressive symptoms indicated by an elevated score (>5) in the Patient Health Care Questionnaire (PHQ-9?) or elevated scores (>9) in the Depression Anxiety and Stress Scale (DASS).
* Elevated Score on Selected questions of the Subchapter "symptoms in the Stomach or Intestines" of the "Rome IV Diagnostic Questionnaire for Adult Functional Gastrointestinal Disorders (Drossman, D. A. (Ed.). (2016). Rome IV: Functional Gastrointestinal Disorders - Disorders of Gut-Brain Interaction (4th ed.). Rome Foundation)

For both arms, the following criteria must be fulfilled:

* Normal or corrected-to-normal vision and hearing.
* Willingness to participate and signed informed consent
* No Medication with cognitive side effects (e.g. psychoactive medications or sleeping pills) or medication affecting gastric motility
* No ectopic heartbeat
* No history of epilepsy or seizure
* No metal implants or devices (e.g. cardiac pacemakers)
* No substance abuse or recent drug consumption
* No pregnancy
* No history of brain- heart- or gastrointestinal surgery
* No skin conditions
* BMI <30

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Heart rate | Pre-stimulation: 25 minutes, stimulation 15 minutes, post-stimulation: 15 minutes
  Objective 1: To improve and validate personalized DLPFC-targeting using a novel HBC-guided frontal mapping technique
  a) Personalization (Study Arm 1, 2): Compare the effects of the HBC protocol (256 sec) between DLPFC sites (Grid-spot versus Beam-F3) versus an active control region (Cz) to induce HBC (within-subjects) and between the three Study Arms (between-subjects). Primary outcome: Change in HR during the HBC-protocol (using the App "Heart Brain Connect").
Heart Rate Variability | Pre-stimulation: 25 minutes, stimulation 15 minutes, post-stimulation: 15 minutes
  Objective 3 (Study Arm 1): To extend HBC-guided rTMS to personalized application of HD-tDCS
  1. Effects of HD-tDCS on the ANS: Compare the pre-post effects of anodal versus sham HD-tDCS (18.75 min) on ANS readouts.
  2. HD-tDCS versus rTMS: Compare the effects of rTMS versus anodal HD-tDCS targeted to the Grid-Spot. Primary outcome: Change in HRV. Secondary outcomes (same): Change in HBC, HR, gut motility, pupil dilation and EDA.

SECONDARY OUTCOMES:
Heart Rate Variability | Pre-stimulation: 25 minutes, stimulation 15 minutes, post-stimulation: 15 minutes
  Objective 2 (Study Arm 1, 2): To explore effects of personalized HBC-guided rTMS on the heart and other ANS measures This hypothesis-generating (exploratory) evaluation will be performed with ANS measures.
  Effects of rTMS on the ANS: Compare the pre-post effects of the Dash protocol (18.75 min) on ANS readouts a) between DLPFC sites (Grid-spot versus Beam-F3) versus an active control region (Cz) (within-subjects) and b) between healthy and symptomatic participants (between-subjects). Primary outcome: Change in HRV
Gut Motility (GM) | Pre-stimulation: 25 minutes, stimulation 15 minutes, post-stimulation: 15 minutes
  Defined as the frequency (cycle time) of contractions within the gastrointestinal tract.
Heart rate | Pre-stimulation: 25 minutes, stimulation 15 minutes, post-stimulation: 15 minutes
  Objective 1: To improve and validate personalized DLPFC-targeting using a novel HBC-guided frontal mapping technique b) Neuroimaging validation (Study Arm 2, 3): Compare DLPFC-sgACC connectivity between DLPFC-sites (Grid-spot versus Beam-F3).
  Primary outcome: Strength of DLPFC-sgACC-anticorrelation.
Pupil dilation | Pre-stimulation: 25 minutes, stimulation 15 minutes, post-stimulation: 15 minutes
  Defined as the expansion of the pupil size (in mm).
Salivary cortisol | 5 minutes (10 minutes before stimulation and 15 minutes after stimulation)
  Defined as the concentration of cortisol hormone present in saliva.
Salivary α-amylase | 5 minutes (10 minutes before stimulation and 15 minutes after stimulation)
  Defined as the enzyme concentration in saliva.
Electrodermal activity (EDA) | Pre-stimulation: 25 minutes, stimulation 15 minutes, post-stimulation: 15 minutes
  Defined as the measure of the electrical conductance of the skin.

CONTACTS AND LOCATIONS:
Overall Officials: Anna-Katharine Brem, PD Dr., Study Chair — University Hospiltal of Old Age Psychiatry and Psychotherapy
Locations (1):
- University Hospital of Old Age Psychiatry and Psychotherapy Bern, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
1. De-identified IPD that underlies the results reported in the publication
  2. After publication of primary results
  3. Open access
  4. Via a data repository following execution of data use agreement
Time Frame: After publication of primary results
Access Criteria: Open access